CLINICAL TRIAL: NCT01352052
Title: Interdisciplinary Rehabilitation and Evaluation Programme for Patients With Chronic Widespread Pain: Randomized Controlled Trial, the IMPROvE Study
Brief Title: Interdisciplinary Rehabilitation of Patients With Chronic Widespread Pain
Acronym: IMPROvE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Frederiksberg University Hospital (Other)
Collaborators: Oak Foundation (Other)
Responsible Party: Principal Investigator, Henning Bliddal, Professor, Frederiksberg University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BDS-2011-099
Record Dates: First submitted 2011-05-04; First posted 2011-05-11 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-08

CONDITIONS: Chronic Widespread Pain; Fibromyalgia
Keywords: chronic widespread pain; fibromyalgia; outcome assessment; functional ability; AMPS; rehabilitation
MeSH Terms: conditions — Chronic Pain; Fibromyalgia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- waiting list assignment (No Intervention): 6 months waiting list assignment followed by the 2-week interdisciplinary rehabilitation programme
- Intervention: interdisciplinary rehabilitation programme (Active Comparator): A two-weeks non-residential, group-based, psycho-educative treatment course conducted by an interdisciplinary team.
  Interventions: Other: interdisciplinary rehabilitation

INTERVENTIONS:
Other: interdisciplinary rehabilitation — A two-weeks non-residential, group-based, psycho-educative, multi-component treatment course conducted by an interdisciplinary team consisting of a rheumatologist, a nurse, occupational therapists, physical therapists, and a psychologist. The rehabilitation Programme comprises of a combination of lectures and group discussions, as well as instructions during physical exercise and task performance. The main focus is on education and adaptations in everyday life. There is a scheduled Programme for every day, with a daily time schedule between four and six hours. There will be a maximum of eight participants in each group.
  Arms: Intervention: interdisciplinary rehabilitation programme

SUMMARY:
The primary objective of the current study is to evaluate the outcome of an interdisciplinary multi-component rehabilitation programme customized to patients with chronic widespread pain (CWP) based on multidimensional diagnostic assessment including sub-grouping, and aiming to improve functional ability in everyday life. The hypothesis is that a patient-focused multi-disciplinary rehabilitation approach will improve both functional ability and quality of life for patients with CWP.

DETAILED DESCRIPTION:
Chronic widespread pain (CWP) is common in the general population and represents a major clinical challenge due to the complexity of the disorder. Apart from pain, CWP comprises a range of secondary features including non-restorative sleep, fatigue, cognitive dysfunction, emotionally distress and disability affecting daily life activities and health-related quality of life. CWP is strongly associated with incapacity for normal employment and poor social participation, and incurs high direct medical costs as well as significant indirect costs, e.g. sick-leave and disability compensation.

Currently there are no official recommendations concerning the diagnosing and management of patients suffering from CWP in the European health care system. The complexity of the condition underlines the necessity of a comprehensive multi-dimensional assessment and a patient-focused multi-component intervention.

The present study is a prospective, pragmatic randomized controlled trial (RCT), with blinded outcome assessors, aiming to evaluate the outcome of an interdisciplinary multi-component rehabilitation programme customized to patients with CWP and focusing on functional ability and adaptations in everyday life. 176 patients with CWP recruited from the department of rheumatology at Frederiksberg Hospital will be consecutively enrolled in the study over a 1-year period. Participants will be randomized to a 2-weeks non-residential, group-based, multi-component treatment course conducted by an interdisciplinary team or 6-months waiting list for the same course.

The instrumentation for intervention planning, as well as for outcome evaluation, will be based on an ICF measurement framework, as recommended by WHO and performance-based assessment of functional ability (AMPS) and self-reported, health-related quality of life (SF-36) will be applied as primary outcome measures.

Overall, the study results is expected to contribute to the development of more cost-effective health care strategies aiming at prevention of mal-adaptive illness behaviour and progressive functional loss in patients suffering from CWP.

ELIGIBILITY:
Inclusion Criteria:

* age above 18
* fulfills the American College of Rheumatology (ACR) 1990 classification criteria of widespread musculoskeletal pain i.e. reporting of pain axially and in all 4 body quadrants for a minimum duration of 3 months
* willing to participate in a 2-week group-based rehabilitation programme

Exclusion Criteria:

* severe physical impairment necessitating assistance in personal activities of daily living
* concurrent history of major psychiatric disorder not related to the pain disorder
* other medical conditions capable of causing patients symptoms (e.g. uncontrolled inflammatory/autoimmune disorder, uncontrolled endocrine disorder, malignancy)
* not Danish speaking
* enrollment in any other clinical trial within the last 30 days

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2011-05; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Assessment of Motor and Process Skills (AMPS) | change from baseline at the end of intervention and 6 months follow-up
  The Assessment of Motor and Process Skills (AMPS) is a performance-based evaluation of ADL ability, developed to establish the extent of an individual's ability to perform and complete daily life tasks independently and in a safe and efficient manner. Further, the AMPS measurement model incorporates the use of Rasch analysis, and therefore provides equal-interval linear measures of the quality of ADL task performances. Two separate measures are reported, one for ADL motor ability (moving self and objects) and one for ADL process ability (organising and adapting actions).
SF-36 Mental Composite Score | change from baseline at the end of intervention and 6 months follow-up

SECONDARY OUTCOMES:
Health related quality of life scales; Short-Form-36 Health Survey (SF-36) | change from baseline at the end of intervention and 6 months follow-up
Disease severity scales;Fibromyalgia Impact Questionnaire (FIQ) | change from baseline at the end of intervention and 6 months follow-up
Anxiety; Generalised Anxiety Disorder (GAD-10) | change from baseline at the end of intervention and 6 months follow-up
Depression; Major Depression Inventory (MDI) | change from baseline at the end of intervention and 6 months follow-up
Pain catastrophizing; Coping Strategy Questionnaire (CSQ) | change from baseline at the end of intervention and at 6 months follow-up
Pain self-efficacy; Pain Self-Efficacy Questionnaire | change from baseline at the end of treatment and at 6 months follow-up
Cognitive functioning; ISPOCD 2 test battery | change from baseline at the end of intervention and 6 months follow-up
Activity intolerance; The Measure of Functional Ability (Tiredness) | change from baseline at the end of intervention and 6 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Bente Danneskiold-Samsøe, Professor, Study Director — The Parker Institute, Frederiksberg University Hospital; Kirstine Amris, MD, Principal Investigator — The Parker Institute, Frederiksberg University Hospital
Locations (2):
- Denmark (2):
  - The Parker Institute, Frederiksberg Hospital, Frederiksberg, Frederiksberg
  - The Parker Institute, Frederiksberg University Hospital, Frederiksberg

REFERENCES:
- [Background] Amris K, Jespersen A, Bliddal H. Self-reported somatosensory symptoms of neuropathic pain in fibromyalgia and chronic widespread pain correlate with tender point count and pressure-pain thresholds. Pain. 2010 Dec;151(3):664-669. doi: 10.1016/j.pain.2010.08.023. Epub 2010 Sep 15. PMID 20832941
- [Background] Waehrens EE, Amris K, Fisher AG. Performance-based assessment of activities of daily living (ADL) ability among women with chronic widespread pain. Pain. 2010 Sep;150(3):535-541. doi: 10.1016/j.pain.2010.06.008. Epub 2010 Jul 3. PMID 20598803
- [Background] Jespersen A, Dreyer L, Kendall S, Graven-Nielsen T, Arendt-Nielsen L, Bliddal H, Danneskiold-Samsoe B. Computerized cuff pressure algometry: A new method to assess deep-tissue hypersensitivity in fibromyalgia. Pain. 2007 Sep;131(1-2):57-62. doi: 10.1016/j.pain.2006.12.012. Epub 2007 Jan 25. PMID 17257757
- See also: Web page of the Parker Institute, Frederiksberg University Hospital, Denmark — http://www.frederiksberghospital.dk/parker